CLINICAL TRIAL: NCT04602481
Title: Living With Primary Ciliary Dyskinesia (Formerly COVID-PCD)
Brief Title: Living With Primary Ciliary Dyskinesia (Living With PCD)
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Selbsthilfegruppe Kartagener Syndrom und Primäre Ciliäre Dyskinesie (Unknown); Verein Kartagener Syndrom und PCD (Unknown); PCD Support UK (Unknown); PCD Foundation (Unknown); PCD Australia (Unknown); European Lung Foundation (Unknown); University of Southampton (Other); Universität Luzern (Other); Associazione Italiana Discinesia Ciliare Primaria Sindrome di Kargagener APS (Unknown); Asociación Nacional de Pacientes con Discinesia Ciliar Primaria (Unknown); Association Dyskinésie Ciliaire Primitive ADCP (Unknown)
Responsible Party: Sponsor
Other Study IDs: Living with PCD (COVID-PCD)
Record Dates: First submitted 2020-10-23; First posted 2020-10-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Living with PCD (formerly COVID-PCD) is a participatory research project that aims to answer emerging questions about primary ciliary dyskinesia (PCD) in order to improve the health and quality of life of people with PCD. Persons with confirmed or suspected PCD from anywhere in the world can participate. The study is advertised through patient support groups and participants register online after they read detailed information about the study. Participants receive a detailed questionnaire when they start the study and a follow-up questionnaire (planned once per year). Occasionally, participants receive extra questionnaires focused on special topics. The study is hosted at the University of Bern and recruitment started on May 30th, 2020.

DETAILED DESCRIPTION:
Background: The study aims to increase knowledge about PCD in order to improve the health and quality of life of people with PCD. The study started in 2020 when PCD patient support groups asked for a study that finds out what happens to people with PCD during the COVID-19 pandemic, because patients with chronic lung disease such as primary ciliary dyskinesia (PCD) were thought to be at increased risk, but no data supported this. PCD patient support groups initiated the idea of a survey that gathers essential knowledge on effects of COVID-19 on people with PCD and makes it available to patients, physicians, and policy makers in real time. After the pandemic, with the continuous encouragement of PCD patient support groups, we want to continue to learn more about other topics important for people living with PCD, such as lung health, mental health or treatment burden by obtaining regular updates via online questionnaires.

Aims: The initial aims of the study was to set up an online surveillance system of COVID-19 for people with PCD. As the aims of the study broaden, we aim to generate knowledge about PCD and study questions raised by people living with PCD and their families. Research questions refer among others to prevalence, severity and progression of disease and symptoms over time, reproductive health, exercise behaviour, nutrition, social and psychological well-being, social inclusion and participation, treatment burden and healthcare related aspects.

Methods: The study population includes all patients with confirmed or suspected PCD from anywhere in the world who can be contacted via patient support groups or find information about the study on the study website. Local support groups invite their contacts using social media and mailing lists. People with PCD can participate via a link on the study website (https://pcd.ispm.ch/en/), where they can read the study information and give consent. Parents of a child with PCD can take part in the study and fill in the study questionnaires with their child. Once registered, participants receive a link via e-mail to the baseline questionnaire with questions about PCD diagnosis, symptoms, and treatment, and health-related behaviours (e.g. exercise), and some general information about the living conditions. Once a year, participants receive a follow-up questionnaire, about current symptoms and treatments to understand who disease progresses with time.

Throughout the study, occasional questionnaires are sent out focusing on emerging questions of interest such as physical activity, mental health, or nutrition. Participants may also suggest topics to be included in these questionnaires and help shape the study. Summaries of results are published on the study website.

Current status: In October 2025, the study received a renewed ethical approval for the renaming to Living with PCD and to cover the broader aims and a wide study re-launch is planned end of 2025. Results from the study, publications, and plain language summaries are listed on the study website (https://pcd.ispm.ch/en/publications/).

ELIGIBILITY:
Inclusion Criteria:

* People of any age with reported suspected or confirmed Primary Ciliary Dyskinesia who gave consent to participate in the study

Exclusion Criteria:

* People who report not to have suspected or confirmed Primary Ciliary Dyskinesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study includes all persons with primary ciliary dyskinesia who can be contacted via patient organisation networks worldwide.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-05-31 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Patient-reported respiratory symptoms | At baseline and through study completion, an average of 1 year
  Prevalence of reported clinical symptoms at different age groups such as cough, shortness of breath, hearing problems
Exercise-behaviour | At baseline and through study completion, an average of 1 year
  Characteristics of exercise-behaviours (frequency, type) at baseline
Treatments | At baseline and through study completion, an average of 1 year
  Information about prescribed treatments for PCD including antibiotics, inhalations, and physiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Claudia E Kuehni, Prof., Principal Investigator — University of Bern; Myrofora Goutaki, Prof, Study Director — University of Bern
Locations (1):
- Institute of Social and Preventive Medicine (ISPM), University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Researchers who wish to use data should submit a concept sheet describing the planned analysis and send it to Prof. Claudia Kuehni (Claudia.kuehni@unibe.ch). The concept sheet will be discussed with the patient advisory group and if agreed, a partial dataset will be prepared by the research team.

REFERENCES:
- [Derived] Schreck LD, Pedersen ESL, Dexter K, Manion M; Living with PCD Study Advisory Group; Massin N, Maitre B, Goutaki M, Kuehni CE. Infertility and pregnancy outcomes among adults with primary ciliary dyskinesia. Hum Reprod Open. 2024 Jun 18;2024(3):hoae039. doi: 10.1093/hropen/hoae039. eCollection 2024. PMID 38962571
- See also: Study website — https://pcd.ispm.ch/en/